CLINICAL TRIAL: NCT00383591
Title: A Phase III, Clinical Trial Comparing the Persistence of GSK Biologicals New Adjuvanted Hepatitis B Vaccine to a Double Dose of Engerix™-B at Months 24, 30, 36, in Pre-haemodialysis/Haemodialysis Patients (≥15 Years of Age)
Brief Title: Comparison of Adjuvanted Hepatitis B Vaccine to Double Dose of Engerix™-B in Pre- /Haemodialysis Patients Aged ≥15 Years
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 208129/047
Record Dates: First submitted 2006-10-02; First posted 2006-10-03 (Estimated); Last update posted 2017-03-23 (Actual); Status verified 2017-03

CONDITIONS: Hepatitis B
MeSH Terms: conditions — Hepatitis B | interventions — Engerix-B

INTERVENTIONS:
Biological: Hepatitis B adjuvanted vaccine
Biological: Engerix-B
  Other Names: Hepatitis B adjuvanted vaccine

SUMMARY:
Persistence of anti-HBs antibodies at Month 24, 30 and 36 in subjects who had completed primary vaccination was evaluated. The anamnestic response to a booster dose was evaluated in subjects with anti-HBs antibody titres < 10 mIU/ml at previous timepoint. The study also evaluated the effect of a booster dose of the vaccine (Month 42) after primary vaccination.

ELIGIBILITY:
Inclusion Criteria:

* Subjects were to have completed primary vaccination course. A male or female > = 15 years of age at the time of the first vaccination.
* Written informed consent obtained from the subject/ from the parents or guardians of the subject.
* If the subject was a female, she was of non-childbearing potential or, if of childbearing potential, she was to be abstinent or use adequate contraceptive precautions for one month prior to enrollment and up to two months after the last vaccination.

Exclusion Criteria:

* Use of any investigational or non-registered drug or vaccine other than the study vaccine within 30 days preceding the booster dose of study vaccine, or planned use during the study period.
* Pregnant or lactating female.

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 120
Dates: Start 2002-03; Study Completion 2004-01 (Actual)

PRIMARY OUTCOMES:
Anti-HBs seroprotection
Response to booster

SECONDARY OUTCOMES:
Solicited, unsolicited symptoms and serious adverse events

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (5):
- GSK Investigational Site, Hradec Králové, Czechia
- GSK Investigational Site, Bandar Tun Razak, Cheras, Malaysia
- Spain (3):
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, Málaga